CLINICAL TRIAL: NCT04789239
Title: OPtimizing Aldosterone Receptor Antagonist Therapy by Sodium Zirconium Cyclosilicate in Heart Failure - Efficacy and Safety of Sodium Zirconium Cyclosilicate in Optimizing Mineralocorticoid Receptor Antagonists Therapy in Heart Failure
Brief Title: OPtimizing Aldosterone Receptor Antagonist Therapy by Sodium Zirconium Cyclosilicate in Heart Failure
Acronym: OPRA-HF
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Michael Fu (Other)
Collaborators: AstraZeneca (Industry); Göteborg University (Other)
Responsible Party: Sponsor-Investigator, Michael Fu, Professor, MD, PhD, FESC, Sahlgrenska University Hospital
Organization: Sahlgrenska University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ESR-19-20262
Record Dates: First submitted 2021-02-25; First posted 2021-03-09 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-04

CONDITIONS: Heart Failure; Hyperkalemia
Keywords: Mineralocorticoid receptor antagonists; Sodium Zirconium Cyclosilicate (SZC); Heart failure with reduced ejection fraction; Treatment
MeSH Terms: conditions — Heart Failure; Hyperkalemia | interventions — sodium zirconium cyclosilicate

STUDY DESIGN:
Intervention Model Description: A multicenter, 1:1 randomized, placebo-controlled, double-blinded study in Sweden of 110 heart failure patients with reduced ejection fraction.
  This study consists of 2 phases: 1) open-label run-in within maximum 2 months, and 2) randomized, double-blinded and placebo-controlled treatment during 6 months.
  The open-label phase, in turn, consists of three periods: run-in (1 - 2 weeks), correction (maximum 72 hours) and maintenance (at least 4 weeks).
  After the open-label run-in phase, upon randomization (1:1 ratio to receive investigational product (IP), either Sodium Zirconium Cyclosilicate (SZC) or placebo, in a blinded manner), SZC will be switched to investigational drug (IP) but with the same dose individually as for SZC before randomization (pre-randomization dose).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: For the 2nd part of study, ie randomized treatment, it is double-blinded with blinding for subjects, endpoint assessors and study personnel. Pharmacy is responsible for masking of differences in appearance, smell and taste, and also packaging and label-ling to ensure blinding.
  Individual treatment codes, indicating the treatment randomisation for each random-ised subject, will be available to Pharmacy where the personnel are independent to the study evaluation.
  The treatment code should not be broken except in medical emergencies when the appropriate management of the subject requires knowledge of the treatment randomisation. The Investigator documents and reports the action to PI, without revealing the treatment given to subject to the PI.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SZC + MRA treated heart failure patients (Experimental): Optimal dose of SZC, which is an approved drug for hyperkalemia in Sweden.
  The subject is treat with 5 mg daily however it can be reduced to once every second day, or inreased to as much as as 10 mg daily, depending on measured potassium levels. This is combined with a mineralcorticoid receptor antagonist (spironolacton or eplerenon), 25 mg or 50 mg depending on what dose they could tolerate.
  Interventions: Drug: Sodium zirconium cyclosilicate
- Placebo + MRA treated heart failure patients (Placebo Comparator): The subject is treat with placebo drug, 5 mg once daily, however it can be reduced to once every second day, or increased to as much as as 10 mg daily, depending on measured potassium levels. This is combined with the dose of mineralcorticoid receptor antagonist (spironolacton or eplerenon) 25 mg or 50 mg depending on what dose they could tolerate.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Sodium zirconium cyclosilicate — SZC is an approved drug in Sweden and subsidized for patients with chronic kidney disease in stages 3 to 5, with or without chronic heart failure, for whom treatment with Resonium is not suitable and for patients with chronic heart failure without con-comitant chronic kidney disease
  Other Names: Lokelma
  Arms: SZC + MRA treated heart failure patients
Other: Placebo — Treatment with the same dose of placebo medicine as they would have received had they been treated with the interventional drug (SZC).
  Arms: Placebo + MRA treated heart failure patients

SUMMARY:
Mineralocorticoid receptor antagonists (MRA) is one of cornerstones in the treatment of heart failure with reduced ejection fraction (HFrEF). However, MRA has been extremely under-used globally. The main reason for this seems to be increased risk of hyperkalemia in individuals on MRA. Theoretically, by limiting the risk of hyperkalemia it could thus be possible to optimize MRA therapy. This is studied in this randomized controlled trial in which it is investigated whethere adding a potassium-binder in combination with MRA treatment prevent hyperkalemia to a greater extent than only using MRA.

The specific aim of this study is to demonstrate the efficacy and safety of Sodium Zirconium Cyclosilicate (SZC) in optimizing MRA in symptomatic patients with HFrEF.

A multicenter, randomized, placebo-controlled, double-blinded study in Sweden (n=110)

The study consists of 2 phases: 1) open-label run-in within maximum 2 months, where all are treated with SZC to test tolarability, and 2) a 1:1 randomized, double-blinded and placebo-controlled treatment during 6 months.

The open-label phase, in turn, consists of three periods: run-in (1 - 2 weeks), correc-tion (maximum 72 hours) and maintenance (4-7 weeks). In addition, post-randomization phase, all patients will be followed by 3 visits (Follow-Up 1, 2 and 3) at 1, 2 and 4 weeks after End of Study (EOS) / End of Treatment (EOT) (which comes first) for further control of kalium and creatinine levels and documentation of current MRA use incl dose.

Sodium Zirconium Cyclosilicate (SZC) (Lokelma)®, 5 g, 10 g, orally, is an approved drug in Sweden. For correction of hyperkalemia, the recommended starting dose is 10 g, three times daily. Once normokalemia has been achieved, the maintenance reg-imen should be started with 5 g once daily. The dose can be titrated up to 10 g once daily or lowered to 5 g once every other day as needed, to maintain a normal level of potassium.

Primary Objective:

To demonstrate the efficacy of Sodium Zirconium Cyclosilicate (SZC) on optimiz-ing MRA in HFrEF, SZC vs Placebo.

Outcome measure: Whether a patient maintains MRA either at a dose ≥ 25 mg daily (for those without MRA at base-line) or a dose increase by 25 mg daily (for those with MRA ≤ 25 mg daily at baseline) and K level in the normal range (3.5-5.0 mmol/L) at the end of study, without rescue therapy due to hy-perkalemia at any point during the randomization phase.

DETAILED DESCRIPTION:
Target subject population

Stable and symptomatic patients with chronic heart failure and LVEF ≤ 40% despite Guideline-Directed Medical Treatment (ACE/ARB/ARNI, beta blockers, SGLT2 inhibitor, MRA) at the discretion of physician´s judgement AND remaining suboptimal treatment of MRA

Duration of treatment

This study consists of 2 treatment phases: 1) Open-label Run-in, and 2) Randomized, pla-cebo-controlled, double-blinded treatment during 6 months. The Open-label phase, in turn, consists of three periods: up-titration (normally 1 - 2 weeks, or longer in some cases), Cor-rection (maximum up to 72 hours) and Maintenance (4-7 weeks)

Investigational product, dosage and mode of administration Sodium Zirconium Cyclosilicate (SZC) (Lokelma)®, 5 g, 10 g, orally, is an approved drug in Sweden. For correction of hyperkalemia, the recommended starting dose is 10 g, three times daily. Once normokalemia has been achieved, the maintenance regimen should be started with 5 g once daily. The dose can be adjusted up to 10 g once daily or lowered to 5 g once every other day as needed, to maintain a normal level of potassium.

ELIGIBILITY:
Inclusion Criteria:

Recruiting will take place mainly from specialist care at University hospitals or Province hospitals in Sweden. But some of patients might have simultaneous follow-up at primary care as well.

Each subject should meet all of the inclusion criteria and none of the exclusion criteria for this study. Under no circumstances can there be exceptions to this rule.

Inclusion criteria

For inclusion in the study subjects should fulfil the following criteria:

1. Obtain signed informed consent prior to any study specific procedures
2. >18 yrs.
3. LVEF ≤ 40% within past 2 years (including recovered EF later on).
4. NYHA II-IV.
5. On optimal treatment including ACE/ARB/ARNI, beta blockers, SGLT2 inhibitor, as per physician´s judgement.
6. Suboptimal treatment with MRA (defined as: no use or ≤ 25 mg daily)
7. And one of following:

   1. Prior hyperkalemia (S-K> 5.0 mmol/L or P-K> 4.8 mmol/L*) during MRA treat-ment within last 24 months, and current S-K ≤ 5.0 or P-K ≤ 4.8 mmol/L
   2. Current S-K 4.5-5.0 mmol/L or P-K 4.3-4.8 mmol/L, and potential risk of hyper-kalemia as indicated by eGFR 30-45 ml/min/1,73 m2 (modified MDRD formula)
   3. Current S-K 5.1-5.9 mmol/L or P-K 4.9-5.7 mmol/L

      * Corresponding plasma K (P-K) level is 0.2 mmol lower than serum K(S-K) (The Nordic Reference Interval Project).

Depending on the S-K status during screening, patients are divided into two groups before treatment initiation /run-in:

* Group 1: Patients who are hyperkalemic (S-K 5.1 - 5.5 mmol/L measured within last 2 weeks)
* Group 2: Patients who are normokalemic (S-K 3.5 - 5.0 mmol/L) during screening but are at a high risk of developing hyperkalemia associated with MRA initiation / increase. Namely, one (or both) of the following:

  * Prescription of MRA within last 12 months and documented hyperkalemia after MRA prescription
  * S-K 4.5-5.0 mmol/L and GFR < 45 mL/min/1,73 m2

Note: All S-K related limits in this protocol concern serum measurements. In Sweden it is plasma that is analyzed, which makes 4.8 mmol/l (plasma) equivalent to 5.0 mmol/L(serum)

Exclusion Criteria:

Subjects should not enter the study if any of the following exclusion criteria are ful-filled:

1. Symptomatic hypotension (< 90/60 mmHg)
2. eGFR < 30 ml/min/1,73 m2 (modified MDRD formula)
3. HF due to restrictive cardiomyopathy, hypertrophic (obstructive) cardio-myopathy or primary valvular disease
4. Current/recent (within 3 months) hospitalization due to myocardial infarc-tion, unstable angina pectoris, coronary revascularization (percutaneous coronary intervention or coronary artery bypass grafting), or other interven-tions (valvular repair/replacement, cardiac transplantation or implantation of a ventricular assistance device)
5. Ongoing or planned dialysis
6. Prior history of hypersensitivity (other than hyperkalemia) to a MRA, or SZC
7. Advanced malignancy requiring treatment
8. History of QT prolongation associated with other medications that required discontinuation of that medication.
9. Congenital long QT syndrome.
10. Symptomatic or uncontrolled atrial fibrillation despite treatment, or asymp-tomatic sustained ventricular tachycardia. Subjects with atrial fibrillation controlled by medication are permitted
11. QTc(f) > 550 msec
12. Currently pregnant (confirmed with positive pregnancy test) or planned pregnancy or breast-feeding
13. Can not sign informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Optimization of MRA usage by Sodium Zirconium Cyclosilicate in HFrEF | 180 days during randomization phase
  Outcome Measure: Whether a patient maintains MRA either at a dose ≥ 25 mg daily (for those without MRA at base-line) or a dose increase by 25 mg daily (for those with MRA ≤ 25 mg daily at baseline) and K level in the normal range (3.5-5.0 mmol/L) at the end of study, without rescue therapy due to hy-perkalemia at any point during the randomization phase.

SECONDARY OUTCOMES:
Maintainance of MRA-dose by Sodium Zirconium Cyclosilicate | 180 days during randomization phase
  Measuring whether a patient is able to maintain at least the same MRA dose at the end of study as at the point of randomization without receiving rescue therapy. SZC vs Placebo
The impact of MRA-optimization on quality of life by Sodium Zirconium Cyclosilicate | 180 days during randomization phase
  Quality of life is measured by KCCQ (the Kansas City Cardiomyopathy Questionnaire): a change in the clinical summary score ( from 0 to 100) with higher scores indicating fewer symptoms and physical limitations, end of study vs at the point of randomizaiton.
The impact of MRA-optimization on symptomatic relief by Sodium Zirconium Cyclosilicate | 180 days during randomization
  Symptomatic relief is evaluated by a composite of change either in NYHA or Lickert Scale as prespecified below:
  1. change in the NYHA functional classifi-cation (I-IV) with higher class indicating more symptomatic and physical limita-tions, or
  2. change in the 5-point Likert scale (5PLS) with higher score indicating the worst possible shortness of breath

OTHER OUTCOMES:
The safety of Sodium Zirconium Cyclosilicate | 180 days during randomization phase
  The difference in safety between two groups is assessed by percent of occurrence of any following prespecified safety endpoints (during the randomization phase):
  1. Patient with S-K <3.0 mmol/l (yes/no)
  2. Patient with S-K ≥6.0 mmol/l (yes/no)
  3. Patient in need of rescue therapy be-cause of hyperkalemia (yes/no)
  4. Patient with fluid retention (general edema, peripheral edema, unrelated to heart failure) (yes/no)
  5. Patient with gastrointestinal events such as constipation, diarrhea, abdominal pain, nausea or vomiting) (yes/no)
  6. Patient with any AE, SAE or DAE (yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Fu, Professor, Principal Investigator — Sahlgrenska University Hospital
Locations (2):
- Sweden (2):
  - Section of Cardiology, Sahlgrenska University Hospital-Östra Hospital, Gothenburg, Västra Götalanddsregion
  - Sahlgrenska University Hospital-Ostra Hospital, Gothenburg

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data with approved ethical permission. All requests will be evaluated but this does not mean all requests will be shared.
Supporting Information: Study Protocol, ICF
Time Frame: We will share the study protocol once a manuscript relating to results of the trial is published in a peer-reviewed medical journal.
Access Criteria: Researchers that ask for access to the study information, were the intention is to evaluate the study and were the anonymity of the study participants is not jeopardized will all be considered for access.